CLINICAL TRIAL: NCT01851863
Title: Compliance With Antidepressant Medication in Treatment of Functional Dyspepsia: A Randomized Comparison of Different Prescribing Behaviors
Brief Title: Compliance With Antidepressant Medication in Treatment of Functional Dyspepsia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Shengliang Chen, professor,chief physician, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RJYYXHNK-001
Record Dates: First submitted 2013-05-04; First posted 2013-05-13 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2014-11

CONDITIONS: Dyspepsia; Compliance; Depression
Keywords: functional dyspepsia; depression; compliance
MeSH Terms: conditions — Dyspepsia; Patient Compliance; Depression | interventions — Omeprazole; Flupenthixol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Flupentixol-Melitracen(psychological and GI) + Omeprazole (Active Comparator): The patients in Group 1 were told that: GI symptoms in FD are attributable to both psychological and GI mechanisms. Flupentixol-Melitracen relieves FD symptoms through both psychological and GI mechanisms.
  Interventions: Drug: Flupentixol-Melitracen(psychological and GI) + Omeprazole
- Flupentixol-Melitracen(psychological) + Omeprazole (Active Comparator): The patients in Group 2 were told that: GI symptoms were attributable to somatization of their psychological problems; and Flupentixol-Melitracen is an antipsychotic drug and primarily acts centrally to alleviate FD symptoms by regulating the psychological condition.
  Interventions: Drug: Flupentixol-Melitracen(psychological) + Omeprazole
- Flupentixol-Melitracen(without explanation) + Omeprazole (Active Comparator): In Group 3, the patients were told only that Flupentixol-Melitrace has been proven to be effective in FD treatment and were not provided additional explanations of the relationships between their GI symptoms and their psychological condition and the reasons for the prescription of Flupentixol-Melitrace.
  Interventions: Drug: Flupentixol-Melitracen(without explanation) + Omeprazole
- proton pump inhibitor (Active Comparator): Prescribe Omeprazole.
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Omeprazole — Prescribe Omeprazole(20mg, po, qd, 30min before breakfast).
  Other Names: Brand name: Aoke (produced by Changzhou Siyao Pharm, China)
  Arms: proton pump inhibitor
Drug: Flupentixol-Melitracen(psychological and GI) + Omeprazole — Prescribe Flupentixol and Melitracen Tablets(one tablet, po, qd, 1 hour after breakfast) and Omeprazole (20mg, po, qd, 30min before breakfast).The patients were told that: GI symptoms in FD are attributable to both psychological and GI mechanisms. Flupentixol-Melitracen relieves FD symptoms through both psychological and GI mechanisms.
  Other Names: Flupentixol and Melitracen Tablets brand name: Deanxit(produced by H.Lundbeck A/S, Copenhagen, Denmark ); Omeprazole brand name: Aoke (produced by Changzhou Siyao Pharm, China)
  Arms: Flupentixol-Melitracen(psychological and GI) + Omeprazole
Drug: Flupentixol-Melitracen(psychological) + Omeprazole — Prescribe Flupentixol and Melitracen Tablets(one tablet, po, qd, 1 hour after breakfast) and Omeprazole (20mg, po, qd, 30min before breakfast). The patients were told that: GI symptoms were attributable to somatization of their psychological problems; and Flupentixol-Melitracen is an antipsychotic drug and primarily acts centrally to alleviate FD symptoms by regulating the psychological condition.
  Other Names: Flupentixol and Melitracen Tablets brand name: Deanxit(produced by H.Lundbeck A/S, Copenhagen, Denmark ); Omeprazole brand name: Aoke (produced by Changzhou Siyao Pharm, China)
  Arms: Flupentixol-Melitracen(psychological) + Omeprazole
Drug: Flupentixol-Melitracen(without explanation) + Omeprazole — Prescribe Flupentixol and Melitracen Tablets(one tablet, po, qd, 1 hour after breakfast) and Omeprazole (20mg, po, qd, 30min before breakfast). The patients were told only that Flupentixol-Melitrace has been proven to be effective in FD treatment and were not provided additional explanations of the relationships between their GI symptoms and their psychological condition and the reasons for the prescription of Flupentixol-Melitrace.
  Other Names: Flupentixol and Melitracen Tablets brand name: Deanxit(produced by H.Lundbeck A/S, Copenhagen, Denmark ); Omeprazole brand name: Aoke (produced by Changzhou Siyao Pharm, China)
  Arms: Flupentixol-Melitracen(without explanation) + Omeprazole

SUMMARY:
The study hypothesis is appropriate clinician-patient communication that provides explanations of the reasons for psychoactive drug prescriptions based on the generation of FD symptoms and the drugs' effects might improve compliance with psychoactive agent regimens among FD patients.

DETAILED DESCRIPTION:
Antidepressive agents have been proved to be effective in the treatment of functional dyspepsia (FD) patients. However, one of the factors that limit therapeutic benefit is the poor compliance with prescribed drugs. The possible reasons for lack of compliance include the patient's health beliefs (e.g., that people who took such agents is possibly considered insane in China), lack of knowledge about antidepressants (that they are addictive or can be stopped on recovery), and aversion to side effects. The investigators propose to examine whether different clinician-patient communication methods could affect adherence to antidepressant drugs in functional dyspepsia patients.

ELIGIBILITY:
Inclusion Criteria:

* met the ROME III criteria for FD;
* education level no lower than high school;
* Hospital Anxiety and Depression Scale (HADS) score > 8 respectively;
* absence of abnormalities in physical examination, laboratory tests (including a routine blood test, blood glucose, and liver function examination), abdominal ultrasonography and upper GI endoscopy within 6 months;
* absence of H. pylori infection

Exclusion Criteria:

* known allergy to omeprazole, flupenthixol or melitracen;
* any evidence of organic digestive diseases;
* reflux-related symptoms only (e.g., retrosternal pain, burning and regurgitation) or predominantly reflux-related symptoms;
* severe psychological symptoms that affected life and work;
* pregnancy or breastfeeding;
* recent myocardial infarction or cardiac arrhythmias;
* previous gastric surgery;
* use of PPIs, psychoactive drugs or other drugs that might affect gastric function within 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shengliang Chen, Study Director — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, China

REFERENCES:
- [Derived] Yan XJ, Li WT, Chen X, Wang EM, Liu Q, Qiu HY, Cao ZJ, Chen SL. Effect of clinician-patient communication on compliance with flupentixol-melitracen in functional dyspepsia patients. World J Gastroenterol. 2015 Apr 21;21(15):4652-9. doi: 10.3748/wjg.v21.i15.4652. PMID 25914475

RESULTS

PARTICIPANT FLOW:
Groups:
- Deanxit(Psychological and GI) + Omeprazole: Prescribe antidepressant drug(Flupentixol and Melitracen Tablets) and proton pump inhibitor(Omeprazole). The patients were told that: GI symptoms in FD are attributable to both psychological and GI mechanisms. Flupentixol-Melitracen relieves FD symptoms through both psychological and GI mechanisms.
- Deanxit(Psychological) + Omeprazole: Prescribe antidepressant drug(Flupentixol and Melitracen Tablets) and proton pump inhibitor(Omeprazole).The patients were told that: GI symptoms were attributable to somatization of their psychological problems; and Flupentixol-Melitracen is an antipsychotic drug and primarily acts centrally to alleviate FD symptoms by regulating the psychological condition.
- Deanxit(Without Explanation) + Omeprazole: Prescribe antidepressant drug(Flupentixol and Melitracen Tablets) and proton pump inhibitor(Omeprazole). The patients were told only that Flupentixol-Melitrace has been proven to be effective in FD treatment and were not provided additional explanations of the relationships between their GI symptoms and their psychological condition and the reasons for the prescription of Flupentixol-Melitrace.
Period: Overall Study
Arm/Group | Deanxit(Psychological and GI) + Omeprazole | Deanxit(Psychological) + Omeprazole | Deanxit(Without Explanation) + Omeprazole | Proton Pump Inhibitor
Started | 65 | 66 | 65 | 66
Completed | 60 | 57 | 60 | 63
Not Completed | 5 | 9 | 5 | 3
Not completed — Did not receive study medication | 2 | 5 | 3 | 0
Not completed — Lost to Follow-up | 3 | 4 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Deanxit(Psychological and GI) + Omeprazole: Prescribe antidepressant drug(Flupentixol and Melitracen Tablets) and proton pump inhibitor(Omeprazole).The patients were told that: GI symptoms in FD are attributable to both psychological and GI mechanisms. Flupentixol-Melitracen relieves FD symptoms through both psychological and GI mechanisms.
- Deanxit(Psychological) + Omeprazole: Prescribe antidepressant drug(Flupentixol and Melitracen Tablets) and proton pump inhibitor(Omeprazole). The patients were told that: GI symptoms were attributable to somatization of their psychological problems; and Flupentixol-Melitracen is an antipsychotic drug and primarily acts centrally to alleviate FD symptoms by regulating the psychological condition.
- Total: Total of all reporting groups
Arm/Group | Deanxit(Psychological and GI) + Omeprazole | Deanxit(Psychological) + Omeprazole | Deanxit(Without Explanation) + Omeprazole | Proton Pump Inhibitor | Total
Number analyzed (Participants) | 65 | 66 | 65 | 66 | 262
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.69 (10.74) | 44.16 (9.26) | 45.72 (10.35) | 46.81 (9.82) | 45.91 (10.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 37 | 35 | 143
  Male | 30 | 30 | 28 | 31 | 119
Region of Enrollment [Number; unit: participants]
  China | 65 | 66 | 65 | 66 | 262

OUTCOME MEASURES:

1. Primary Outcome: Compliance of Flupentixol-Melitracen
Description: The patients were asked to keep a diary to record their medication intake. At each visit (weeks 1, 2, 4, 8), the patient bring back the drug bottle and the diary, then the physician recorded the number of pills remaining in the bottle. Pills remained more than 20% at any visit or seven days of consecutive abstinence were adopted as the criterion for identifying therapy noncompliance.
Time Frame: weeks 1, 2, 4, 8
Measure: Number; unit: participants
Arm/Group | Deanxit(Psychological and GI) + Omeprazole | Deanxit(Psychological) + Omeprazole | Deanxit(Without Explanation) + Omeprazole
Number analyzed (Participants) | 65 | 66 | 65
participants | 44 | 28 | 31

2. Secondary Outcome: Change From Baseline in Dyspepsia Symptom Questionnaire at Week 8
Description: The severity of patients' dyspeptic symptoms were assessed using the Leeds Dyspepsia Questionnaire (LDQ) at week 0 and 8. The LDQ contains eight items about epigastric pain, retro-sternal pain, regurgitation, nausea, vomiting, belching, early satiety and dysphagia with six grades for each item and a sum of the eight symptom scores make the LDQ score.LDQ scores of 0 - 4 were classified as very mild dyspepsia, 4 - 8 as mild dyspepsia, 9 -15 as moderate dyspepsia, and > 15 as severe or very severe dyspepsia. The change of LDQ scores was calculated by LDQ scores of 8 weeks minus baseline, with lower values represent a better outcome.
Time Frame: week 0 and 8
Measure: Mean (Full Range); unit: units on LDQ scale
Groups:
- Deanxit(Psychological and GI) + Omeprazole: Prescribe antidepressant drug(Flupentixol and Melitracen Tablets) and proton pump inhibitor(Omeprazole) .The patients were told that: GI symptoms in FD are attributable to both psychological and GI mechanisms. Flupentixol-Melitracen relieves FD symptoms through both psychological and GI mechanisms.
Arm/Group | Deanxit(Psychological and GI) + Omeprazole | Deanxit(Psychological) + Omeprazole | Deanxit(Without Explanation) + Omeprazole | Proton Pump Inhibitor
Number analyzed (Participants) | 60 | 57 | 60 | 63
units on LDQ scale | -3.85 [-9 to 2] | -2.51 [-8 to 3] | -2.49 [-6 to 3] | -1.31 [-7 to 2]

3. Secondary Outcome: Change From Baseline in Psychiatric Symptom on Hospital Anxiety and Depression Scale at Week 8
Description: Each patient was surveyed using the Hospital Anxiety and Depression Scale to assess the psychiatric symptom at week 0 and 8.The HADS consists of 14 items, seven of which assess anxiety, and seven assess depression. The anxiety and depression subscales were calculated independently. The patients were asked to answer each item on a four-point (0 - 3) scale. Scores of 0 to 7 on either subscale can be regarded as within the normal range, scores of 8 to 10 are suggestive of the presence of the respective state, and scores of 11 or higher indicate the probable presence of the respective mood disorder. The change of HADS scores was calculated by HADS anxiety and depression scores of 8 weeks minus baseline, with lower values indicate better outcome.
Time Frame: week 0 and 8
Measure: Mean (Full Range); unit: units on HADS score
Arm/Group | Deanxit(Psychological and GI) + Omeprazole | Deanxit(Psychological) + Omeprazole | Deanxit(Without Explanation) + Omeprazole | Proton Pump Inhibitor
Number analyzed (Participants) | 60 | 57 | 60 | 63
units on HADS score
  HADS anxiety score | -4.46 [-12 to 3] | -2.29 [-9 to 3] | -2.78 [-9 to 4] | -1.68 [-6 to 3]
  HADS depression score | -4.82 [-10 to 2] | -2.25 [-7 to 5] | -2.86 [-9 to 4] | -1.88 [-6 to 5]

4. Other Pre Specified Outcome: Number of Participants With Adverse Reaction
Description: Number of participants with adverse reactions were recorded to analyze the safety profile of treatment.
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Deanxit(Psychological and GI) + Omeprazole | Deanxit(Psychological) + Omeprazole | Deanxit(Without Explanation) + Omeprazole | Proton Pump Inhibitor
Number analyzed (Participants) | 60 | 57 | 60 | 63
participants | 6 | 9 | 5 | 2

ADVERSE EVENTS:
Arm/Group | Deanxit(Psychological and GI) + Omeprazole | Deanxit(Psychological) + Omeprazole | Deanxit(Without Explanation) + Omeprazole | Proton Pump Inhibitor
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/66 | 0/65 | 0/66
Other Adverse Events (participants affected / at risk) | 6/65 | 9/66 | 5/65 | 2/66
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deanxit(Psychological and GI) + Omeprazole (N=65) | Deanxit(Psychological) + Omeprazole (N=66) | Deanxit(Without Explanation) + Omeprazole (N=65) | Proton Pump Inhibitor (N=66)
Insomnia (Nervous system disorders) | 3 | 4 | 4 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Dry mouth (General disorders) | 1 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Skin rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No